CLINICAL TRIAL: NCT07345819
Title: Dexamethasone vs. Placebo in Children and Youth Hospitalized for Orbital Cellulitis: the VISION Pilot Randomized Clinical Trial
Brief Title: Dexamethasone vs. Placebo in Children and Youth Hospitalized for Orbital Cellulitis
Acronym: VISION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Peter Gill, Staff Paediatrician and Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3800
Record Dates: First submitted 2026-01-06; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Orbital Cellulitis
Keywords: orbital cellulitis; pilot trial; pilot RCT; preseptal cellulitis; periorbital cellulitis; dexamethasone; corticosteroid; inpatient; RCT; randomized controlled trial; pediatric; paediatric; children; youth
MeSH Terms: conditions — Orbital Cellulitis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Dexamethasone 0.3 mg/kg (max dose 12 mg) IV after randomization, and a second dose 24 hours (+/-8 hours) after the first dose
  Interventions: Drug: Dexamethasone 0.3mg/kg
- Placebo (Placebo Comparator): Sodium Chloride 0.9% IV after randomization and second dose 24 hours (+/- 8 hours) after the first dose
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Dexamethasone 0.3mg/kg — SANDOZ-DEXAMETHASONE SODIUM PHOSPHATE INJ USP 4MG/ML (5 mL vial) (DIN# 00664227) or any brand available commercially in the Canadian market.
  Dexamethasone 0.3 mg/kg (max dose 12 mg) will be given by IV after randomization. The second dose will be given 24 hours (+/-8 hours) after the first dose. The most recent weight recorded in the patient's chart will be used for the dose calculation.
  Arms: Intervention
Drug: Placebo Control — Sodium Chloride 0.9% Injection USP Placebo Baxter brand (or any commercially available in the Canadian market) given by IV, first dose administered after randomization and second dose 24 hours (+/- 8 hours) after the first.
  Arms: Placebo

SUMMARY:
The goal of this pilot randomized controlled trial is to understand whether we can successfully conduct a larger definitive clinical trial in the future. The current pilot study will test various aspects of the larger trial and help us improve its design if needed. The investigators are mainly interested in knowing whether they can (1) recruit enough patients, (2) administer the intervention, and (3) collect all the data needed from patients. The definitive randomized controlled trial will assess if dexamethasone is superior to placebo for treating children and youth hospitalized with orbital cellulitis.

DETAILED DESCRIPTION:
This is a double-blinded, placebo-controlled, internal pilot randomized controlled trial, with two parallel groups with a 1:1 allocation ratio, at The Hospital for Sick Children (Toronto, ON) and Stollery Children's Hospital (Edmonton, AB).The purpose of the study is to determine the feasibility of a definitive randomized controlled trial, which will determine whether IV dexamethasone 0.3 mg/kg after randomization and 24 hours later (2 doses total) is superior to placebo for children and youth hospitalized with orbital cellulitis.

Children and youth (n=30) hospitalized with orbital cellulitis will be randomized to receive IV dexamethasone 0.3 mg/kg (first dose after randomization, second dose 24 hours later) or placebo. The primary feasibility outcome of this pilot trial is recruitment rate. Secondary feasibility outcomes include (a) intervention fidelity, (b) completion of definitive trial primary, and (c) completion of definitive trial secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2.00 months -17.99 years (prior to 18th birthday)
2. Confirmed or suspected diagnosis of orbital cellulitis as determined by the attending physician, medical team, and/or delegate's clinical judgement, based on one or more features of orbital cellulitis (i.e., ophthalmoplegia, pain and/or limitation with extraocular movements, chemosis, blurred vision, eye swollen shut, and/or proptosis).
3. Scheduled to be admitted or admitted to hospital for less than 36 hours.
4. Informed consent provided in accordance with institutional policies

Exclusion Criteria:

1. Transferred directly from outside hospital inpatient setting to a participating hospital site's inpatient setting with over 36 hours having passed since admission to outside hospital. If within 36 hours, patient is eligible.
2. Treatment with IV or PO systemic corticosteroids within 1 week of presentation
3. Recent hospital admission for orbital cellulitis within 1 week of presentation
4. Current systemic fungal infection
5. Contraindication for dexamethasone or components of dexamethasone IV formulation
6. Clinically relevant varicella exposure in the previous 21 days
7. Previous enrollment in this study
8. No telephone/mobile/email
9. Poor mastery of English, or medical interpreter not available for languages other than English

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From start of recruitment to end of recruitment (anticipated 18 months).
  Recruitment rate is measured as the number of patients agreeing to participate in the trial and are randomized, divided by the number of patients screened as eligible at 18 months after initiation of the trial recruitment (per site).

SECONDARY OUTCOMES:
Intervention fidelity | 96 hours after the patient is admitted to hospital.
  Intervention fidelity is the proportion of randomized patients who receive the intervention or placebo at the correct dose and time, without receiving any off-protocol corticosteroids, at each site. It will be assessed 96 hours after hospital admission, defined as the patient receiving two doses of 0.3 mg/kg dexamethasone or placebo (first dose after randomization; second dose at 24 +/- 8hrs after first dose).
Completion of definitive trial primary and secondary outcomes | Three months after the patient is discharged from hospital.
  Completion of definitive trial primary and secondary outcomes is defined as the proportion of randomized patients with complete data for the definitive trial primary outcome (length of hospital stay) and the definitive trial secondary outcomes, at each site.
  The definitive trial secondary outcomes include: Surgical intervention, clinical outcomes (e.g. vision, pain, swelling), healthcare use (ICU admission, revisits to medical care and hospital), perceived stress experienced by parents, and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Gill, MD, DPhil, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Stollery Children's Hospital, Edmonton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonsalves CL, Borkhoff C, Mahant S, Drouin O, Pound C, Quet J, Wahi G, Bayliss A, Vomiero G, Foulds JL, Kanani R, Sakran M, Sehgal A, Pullenayegum E, Widjaja E, Reginald A, Wolter NE, Parkin PC, Gill PJ; Periorbital and Orbital Cellulitis (POC) Multicentre Study Group and Canadian Paediatric Inpatient Research Network (PIRN). Association of systemic corticosteroids and clinical outcomes in children hospitalised with severe orbital infections. BMJ Paediatr Open. 2025 Dec 11;9(1):e004161. doi: 10.1136/bmjpo-2025-004161. PMID 41381246
- [Background] Kornelsen E, Mahant S, Parkin P, Ren LY, Reginald YA, Shah SS, Gill PJ. Corticosteroids for periorbital and orbital cellulitis. Cochrane Database Syst Rev. 2021 Apr 28;4(4):CD013535. doi: 10.1002/14651858.CD013535.pub2. PMID 33908631
- [Background] Gill PJ, Mahant S, Hall M, Parkin PC, Shah SS, Wolter NE, Mestre M, Markham JL. Association Between Corticosteroids and Outcomes in Children Hospitalized With Orbital Cellulitis. Hosp Pediatr. 2022 Jan 1;12(1):70-89. doi: 10.1542/hpeds.2021-005910. PMID 34877598